CLINICAL TRIAL: NCT03343470
Title: The Observational Prospective Multicentric Study on Melatonin and Cortisol Circadian Rhythm in CusHing SyndrOme Patients in Active Phase and dUring RemiSsion.
Brief Title: The Circadian Rhythm in CusHing SyndrOme in Active Phase and dUring RemiSsion (TheHOURS)
Acronym: TheHOURS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Federico II University (Other); University of Palermo (Other); University of Florence (Other); Ospedali Riuniti Ancona (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Assistant Professor, University of Roma La Sapienza
Other Study IDs: Adrenal_2
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Cushing Syndrome
Keywords: Cushing Syndrome; Adrenal Insufficiency; Peripheral blood mononuclear cells; Melatonin; Cortisol; Immunological profile; Cushing Disease
MeSH Terms: conditions — Cushing Syndrome; Adrenal Insufficiency; Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cushing Syndrome (active phase): Patients displaying biochemical and clinical features of active Cushing's syndrome
- Cushing Syndrome (during remission): Patients at 3-6 months from remission with cortisol levels in the normal range

SUMMARY:
This is an observational, open, prospective multi-centre study designed to evaluate melatonin and cortisol circadian rhythm, immunological profile and anthropometric parameters in Cushing Syndrome patients during active Remission state.

DETAILED DESCRIPTION:
Cushing Syndrome is a severe condition caused by prolonged exposure to high levels of glucocorticoids.

This is a disease with high morbidity and mortality due to metabolic, cardiovascular, coagulative, psychiatric complications of hypercortisolism.

The loss of circadian secretion of cortisol is one of the most sensitive and specific diagnostic features of Cushing's Syndrome that normalizes during remission. The evaluation of the circadian rhythm of cortisol is one of the diagnostic tests recommended by the guidelines to evaluate the state of the disease's activity.

Studies in literature have shown several correlations between states of hypercortisolism and circadian secretion of melatonin, displaying reduced melatonin secretion throughout the day and the suppression of circadian rhythm of cortisol. However, the dynamics of the normalization of melatonin circadian rhythm during remission from Cushing syndrome are unclear.

Therefore, the aim of our study is to evaluate the changes in circadian secretion of melatonin in Cushing's syndrome during active disease and during remission (3 and 6 months), according to the rational scientific influence of endogenous hypercortisolism on the function of the pineal gland. In addition, the changes in circadian secretion of cortisol, of mononuclear cells of the blood (PBMC) and of anthropometric-metabolic parameters, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Cushing Syndrome during active phase

Exclusion Criteria:

* Malignancy
* Alcoholism or drug addiction
* Psychiatric disorders
* Clinical or laboratory signs of significant cardiovascular, hepatobiliary disease
* Clinically significant renal dysfunction
* Pregnancy
* Any medication with agents which could interfere with glucocorticoid kinetics and melatonin secretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cushing Syndrome patients in active phase and during remission at 3 and 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in measurement of melatonin secretion at 3 and 6 months | 0, +3 months, +6 months
  single outcome measurement of melatonin secretion

SECONDARY OUTCOMES:
Evaluation of immunological profile at baseline, 3 and 6 months | 0, +3 months, +6 months
  composite outcome measure consisting of simultaneous measurement of: PBMC profiling with flow cytometry, Full count blood cell
Evaluation of cortisol circadian rhythm | 0, +3 months, +6 months
  single outcome measure of circadian cortisol secretion
Change from baseline in measurement of anthropometric-metabolic parameters at 3 and 6 months | 0, +3 months, +6 months
  composite outcome measure consisting of simultaneous measurement of:body weight (kg), waist circumference (cm), blood pressure and pulse

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — Dept. Experimental Medicine
Locations (1):
- Department of Experimental Medicine, Rome, Italy

REFERENCES:
- [Result] Tomova A, Kumanov P, Robeva R, Manchev S, Konakchieva R. Melatonin secretion and non-specific immune responses are differentially expressed in corticotropin-dependent and corticotropin-independent Cushing's syndrome. Med Sci Monit. 2008 Jun;14(6):CR327-332. PMID 18509277
- [Result] Pivonello R, De Leo M, Cozzolino A, Colao A. The Treatment of Cushing's Disease. Endocr Rev. 2015 Aug;36(4):385-486. doi: 10.1210/er.2013-1048. Epub 2015 Jun 11. PMID 26067718
- [Result] Piovesan A, Terzolo M, Borretta G, Torta M, Buniva T, Osella G, Paccotti P, Angeli A. Circadian profile of serum melatonin in Cushing's disease and acromegaly. Chronobiol Int. 1990;7(3):259-61. doi: 10.3109/07420529009056984. PMID 2268888
- [Result] Fevre-Montange M, Tourniaire J, Estour B, Bajard L. 24 hour melatonin secretory pattern in Cushing's syndrome. Clin Endocrinol (Oxf). 1983 Aug;19(2):175-81. doi: 10.1111/j.1365-2265.1983.tb02979.x. PMID 6684004
- [Result] Angeli A, Gatti G, Sartori ML, Masera RG. Chronobiological aspects of the neuroendocrine-immune network. Regulation of human natural killer (NK) cell activity as a model. Chronobiologia. 1992 Jul-Dec;19(3-4):93-110. No abstract available. PMID 1478121